CLINICAL TRIAL: NCT00167362
Title: Rehabilitation, Brain Function and Early Schizophrenia
Brief Title: Cognitive Enhancement Therapy for Early-Stage Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Matcheri S. Keshavan MD, PI, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH060902 (NIH); R01MH060902 (NIH); DATR A2-AISZ
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognition; Enhancement; Randomized
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive cognitive enhancement therapy
  Interventions: Behavioral: Cognitive enhancement therapy (CET)
- 2 (Placebo Comparator): Participants will receive enriched supportive therapy
  Interventions: Behavioral: Enriched supportive therapy (EST)

INTERVENTIONS:
Behavioral: Cognitive enhancement therapy (CET) — Using 80 to 100 hours of graduated exercises in computer assisted training, coupled with structured but unrehearsed in vivo social group interactions, CET tries to shift an early developmental reliance on effortful, serial and verbatim cognitive processing to a more gistful, less effortful and spontaneous abstraction of social themes. CET uses attention, memory and problem solving software from three exercises from Ben-Yishay's Orientation Remediation Module (the Attention Reaction Conditioner, Zero Accuracy Conditioner, and Time Estimates) that are graduated in difficulty and designed to enhance vigilance, selective attention, the ability to shift between auditory and visual modalities, and rapid decision-making.
  Arms: 1
Behavioral: Enriched supportive therapy (EST) — EST is the commonly recommended (Spaulding 1992) treatment for control and experimental subjects in psychosocial trials. EST is a two-staged treatment that requires weekly one-hour sessions in Phase 1 and biweekly sessions in Phase 2. Some practice principles (e.g., psychoeducation and relaxation training) are provided during the group exercises for CET patients, but individually for EST patients. No attempt is made to control for hours of contact between EST and CET, since offering three hours of supportive therapy to EST subjects is neither logistically feasible nor faithful to the goals and methods of supportive therapy. Further, neurobiological hypotheses related to treatment specificity would be best tested by clear differences in treatment intensity and content.
  Arms: 2

SUMMARY:
This study will determine the effectiveness of cognitive enhancement therapy (CET) in treating cognitive abnormalities in people experiencing the early stages of schizophrenia.

DETAILED DESCRIPTION:
In this study, we wish to determine the neurobiological predictors and the relative efficacy of Cognitive Enhancement Therapy (CET) in ameliorating specific cognitive abnormalities presumably mediated by PFC and related brain structures, among younger, early-course schizophrenia patients who potentially have a better prognosis. A series of recent-onset schizophrenic patients, whose psychotic symptoms have successfully been stabilized on an atypical antipsychotic drug for one year following initiation of treatment, will be randomized to CET combined with an enriched supportive therapy (EST) or EST alone, and treated for two years. Subjects will have been assessed on neurobehavioral and clinical indices immediately prior to beginning CET or EST (corresponding with the CNMD 1-year follow-up) and in the proposed study will again be assessed after 1 and 2 years of psychosocial treatment. In a smaller subset of patients, we will also seek to collect preliminary data on the efficacy of CET in reversing the neurobiological alterations in the PFC. The hypotheses of this study are:

1. The presence of relatively well preserved PFC structure and function (PFC volume, activation with fMRI, and metabolism as measured by proton MRS) at baseline will predict a better response to CET (Neurobiological Prediction Hypothesis).
2. CET combined with "enriched" supportive psychotherapy (EST) will be more effective than EST alone in ameliorating social and non-social cognitive deficits of patients with early schizophrenic illness whose psychotic symptoms have been stabilized on maintenance chemotherapy (The Treatment Efficacy Hypothesis).
3. CET will result in additive, positive effects on neurocognitive parameters that were not observed following one year of antipsychotic medication, using a "sequential" treatment design in a subset of patients in whom we have pre-neuroleptic baseline data from CNMD studies (The Treatment Specificity Hypothesis).

Study Design: Subjects will be randomly assigned, once stabilized clinically, to CET plus EST (n = 30) or EST alone (n = 30) and then treated for up to two years. Clinical, neuropsychological, neurological and functional neuroimaging assessments will be administered at baseline and at two annual follow-ups. At the end of CET or EST treatment, subjects will be asked to come back quarterly to meet informally with either their Cognitive Enhancement Therapy clinicians and former group members, or with their Enriched Supportive Therapy clinician. The purpose of these visits is for us to learn more about the successes that patients have had, or about the difficulties that they might have had since leaving the program. Clinician(s) will also share information obtained during this follow-up which might help patient in overcoming these difficulties. At the end of the one-year period post EST or CET treatment, subjects will be assessed on all measures, except for diagnostic, imaging and blood studies.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia, schizoaffective or schizophreniform disorder at the time of initial assessment
* Pre-treatment illness duration an average of 5 years, not to exceed 8 years
* Stable positive symptoms (e.g., if present do not grossly interfere with behavior such as command hallucinations or delusions)
* Currently maintained and compliant with prescribed antipsychotic medication
* Socially and cognitively disabled, e.g., meet criteria on a Cognitive Style Scale (score greater than or equal to 7), and Social Cognition Disability Scale (score greater than or equal to 12).

Exclusion Criteria:

* Alcohol/drug abuse or dependence that has significantly interfered with adjustment in the past two months (e.g., patients currently undergoing D and A treatment must successfully complete their recovery program prior to referral)
* Organic brain syndrome, including HIV illness (due to its effect on CNS function)
* IQ below 80 or language skills below the sixth grade level
* Medical contraindications that preclude an appropriate antipsychotic medication
* Persistent suicidality

Ages: 16 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2001-08; Primary Completion 2009-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Clinical, neuropsychological, and functional outcomes | Measured at Years 1 and 3

SECONDARY OUTCOMES:
Neuroimaging parameters | Measured at Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Matcheri S Keshavan, MD, Principal Investigator — University of Pittsburgh; Gerard E Hogarty, MSW, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Hogarty GE. Reinventing evidence-based interventions? Psychiatr Serv. 2005 Sep;56(9):1156; author reply 1156-7. doi: 10.1176/appi.ps.56.9.1156. No abstract available. PMID 16148337
- [Background] Hogarty GE, Flesher S, Ulrich R, Carter M, Greenwald D, Pogue-Geile M, Kechavan M, Cooley S, DiBarry AL, Garrett A, Parepally H, Zoretich R. Cognitive enhancement therapy for schizophrenia: effects of a 2-year randomized trial on cognition and behavior. Arch Gen Psychiatry. 2004 Sep;61(9):866-76. doi: 10.1001/archpsyc.61.9.866. PMID 15351765
- [Background] Hogarty GE. Medication adherence studies in schizophrenia. Am J Psychiatry. 2004 Mar;161(3):581-2; author reply 582-3. doi: 10.1176/appi.ajp.161.3.581-a. No abstract available. PMID 14992994
- [Background] Hogarty GE. Cognitive rehabilitation of schizophrenia. Harv Ment Health Lett. 2000 Aug;17(2):4-6. No abstract available. PMID 10927651
- [Background] Hogarty GE, Flesher S. Practice principles of cognitive enhancement therapy for schizophrenia. Schizophr Bull. 1999;25(4):693-708. doi: 10.1093/oxfordjournals.schbul.a033411. PMID 10667740
- [Background] Keshavan MS, Hogarty GE. Brain maturational processes and delayed onset in schizophrenia. Dev Psychopathol. 1999 Summer;11(3):525-43. doi: 10.1017/s0954579499002199. PMID 10532623
- [Background] Hogarty GE, Ulrich RF. The limitations of antipsychotic medication on schizophrenia relapse and adjustment and the contributions of psychosocial treatment. J Psychiatr Res. 1998 May-Aug;32(3-4):243-50. doi: 10.1016/s0022-3956(97)00013-7. PMID 9793877
- [Derived] Eack SM, Hogarty GE, Cho RY, Prasad KM, Greenwald DP, Hogarty SS, Keshavan MS. Neuroprotective effects of cognitive enhancement therapy against gray matter loss in early schizophrenia: results from a 2-year randomized controlled trial. Arch Gen Psychiatry. 2010 Jul;67(7):674-82. doi: 10.1001/archgenpsychiatry.2010.63. Epub 2010 May 3. PMID 20439824